CLINICAL TRIAL: NCT02236507
Title: Evaluation of Anorectal Area in Children Using 3D High Resolution Anorectal Manometry.
Brief Title: Normal Values for 3D High Resolution Anorectal Manometry in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Marcin Banasiuk, MD, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Banasiuk2014 A
Record Dates: First submitted 2014-08-31; First posted 2014-09-10 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Children; Anorectal Disorder
MeSH Terms: conditions — Rectal Diseases

ARMS (1):
- children without anorectal disorders (Other): All children will be investigated by 3D high resolution anorectal manometry procedure
  Interventions: Device: 3D high resolution anorectal manometry

INTERVENTIONS:
Device: 3D high resolution anorectal manometry — Procedure will take about 15 min. During procedure resting, voluntary squeeze, bear down maneuver, cough reflex, ano-anal reflex and Rectoanal Inhibitory Reflex will be obtained, if possible.

SUMMARY:
Anorectal 3D high resolution manometry (3D HRM) is the most advanced version of manometry equipment and has been recently introduced into clinical practice. It is the most precise method to assess the anal sphincter pressure function and may be crucial for planning and controlling surgical procedures of the anorectal area. Normal values in pediatric population have not been established.

The aim of this study is complex evaluation of anorectal function in children without symptoms from lower GI tract and establishment of normal values.

ELIGIBILITY:
Inclusion Criteria:

* parental agreement
* age: 1 to 18 yr

Exclusion Criteria:

* parental disagreement
* children younger than 1 yr
* children after the surgery for anorectal malformations
* children with constipation during the last 10 months
* children with nonretentive fecal soiling
* children with inflammatory bowel diseases or any other type of large bowel inflammation
* children with anal fissure, anal varices, inflammation of the anorectal area or any other disease that may interfere with function of anorectum

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mean and maximum sphincters pressures during rest, voluntary squeeze and bear down maneuvers and Asymmetry of the anal canal | up to 20 minutes
  Pressures during voluntary maneuvers will be obtained if cooperation with a child will be possible

SECONDARY OUTCOMES:
Presence of Rectoanal Inhibitory Reflex | up to 5 minutes
  Amount of air in a balloon needed to elicit Rectoanal Inhibitory Reflex
Presence of dyssynergic defecation | up to 1 minute
  Percent of children without constipation but with dyssynergic defecation pattern
Presence of Cough Reflex | 10 seconds
Presence of Ano-anal Reflex | 10 seconds
Presence of discomfort during the procedure | up to 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Banasiuk, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of Pediatric Gastroenterology and Nutrition, Warsaw, Poland

REFERENCES:
- [Derived] Banasiuk M, Banaszkiewicz A, Dziekiewicz M, Zaleski A, Albrecht P. Values From Three-dimensional High-resolution Anorectal Manometry Analysis of Children Without Lower Gastrointestinal Symptoms. Clin Gastroenterol Hepatol. 2016 Jul;14(7):993-1000.e3. doi: 10.1016/j.cgh.2016.01.008. Epub 2016 Jan 25. PMID 26820403